CLINICAL TRIAL: NCT00915863
Title: A Prospective Randomized Controlled Trial Comparing Isolated Roux-en-Y Reconstruction With Billroth-II-type Reconstruction After Pancreaticoduodenectomy
Brief Title: Evaluation of Isolated Roux-en-Y Reconstruction After Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP-0901
Record Dates: First submitted 2009-05-22; First posted 2009-06-08 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Pancreatic Neoplasms; Bile Duct Neoplasms; Ampullary Neoplasms; Duodenal Neoplasms; Pancreatitis
Keywords: pancreaticoduodenectomy; pancreatic fistula; reconstruction; isolated Roux-en-Y
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms; Duodenal Neoplasms; Pancreatitis; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Billroth-II-type (Active Comparator): Billroth-II-type reconstruction after pancreaticoduodenectomy
  Interventions: Procedure: Billroth-II-type reconstruction
- Isolated Roux-en-Y (Experimental): Isolated Roux-en-Y type reconstruction after pancreaticoduodenectomy
  Interventions: Procedure: Isolated Roux-en-Y type reconstruction

INTERVENTIONS:
Procedure: Billroth-II-type reconstruction — surgical procedure
  Other Names: Child reconstruction
  Arms: Billroth-II-type
Procedure: Isolated Roux-en-Y type reconstruction — surgical procedure
  Other Names: Roux-en-Y reconstruction
  Arms: Isolated Roux-en-Y

SUMMARY:
The purpose of this study is to evaluate the incidence of complications with the isolated Roux-en-Y reconstruction after pancreaticoduodenectomy in pancreatic tumor and periampullary tumor patients. A prospective randomized controlled trial was conducted to compare the incidence of complications with isolated Roux-en-Y reconstruction with those of Billroth-II-type reconstruction after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
The purpose of this study is to clarify whether isolated Roux-en-Y reconstruction declines the incidence of postoperative complications after pancreaticoduodenectomy compared with Billroth-II-type reconstruction. Especially, it is important to decline the incidence of pancreatic fistula, because pancreatic fistula affects a postoperative course. However, there is no report that demonstrated postoperative complications of isolated Roux-en-Y compared with those of Billroth-II-type reconstruction. We conducted a prospective randomized trial on patients who underwent pancreaticoduodenectomy.

Patients with pancreatico-biliary disease who were performed pancreaticoduodenectomy at Wakayama Medical University Hospital.

The primary endpoint was defined as the incidence of pancreatic fistula. The secondary endpoints were the incidence of other postoperative complications, mortality, delayed gastric emptying, intra-abdominal hemorrhage, and intra-abdominal abscess. Patients were recruited into this study before surgery, on the basis of whether pancreatic head resection was anticipated at Wakayama Medical University Hospital (WMUH) for pancreatic head and periampullary disease, and appropriate informed consent was obtained. Exclusion criteria was 1) young patients (less than 20-year-old), 2) patients with severe complications which were possible to prolong hospital stay, 3) patients undergone hemodialysis, 4) patients combined resection of other organs, 5) patients who were diagnosed inadequacy for this study by a physician, and 6) patients without an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* the patients had undergone pancreatic head resection at Wakayama Medical University the patients obtained appropriate informed consent

Exclusion Criteria:

* young patients (less than 20-years-old)
* patients with severe complications which were possible to prolong hospital stay
* patients undergone hemodialysis
* patients combined resection of other organs
* patients who were diagnosed inadequacy for this study by a physician
* patients without an informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-10 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
the incidence of pancreatic fistula | 3 months after operation

SECONDARY OUTCOMES:
the incidence of other postoperative complications, mortality, delayed gastric emptying, intra-abdominal hemorrhage, and intra-abdominal abscess | 3 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Masaji Tani, MD, Study Chair — Wakayama Medical University
Locations (1):
- Wakayama Medical University , Second Department of Surgery, 811-1 Kimiidera, Wakayama, Wakayama, Japan

REFERENCES:
- [Background] Kawai M, Tani M, Terasawa H, Ina S, Hirono S, Nishioka R, Miyazawa M, Uchiyama K, Yamaue H. Early removal of prophylactic drains reduces the risk of intra-abdominal infections in patients with pancreatic head resection: prospective study for 104 consecutive patients. Ann Surg. 2006 Jul;244(1):1-7. doi: 10.1097/01.sla.0000218077.14035.a6. PMID 16794381
- [Background] Tani M, Kawai M, Terasawa H, Ina S, Hirono S, Uchiyama K, Yamaue H. Does postoperative chemotherapy have a survival benefit for patients with pancreatic cancer? J Surg Oncol. 2006 May 1;93(6):485-90. doi: 10.1002/jso.20440. PMID 16615151
- [Background] Tani M, Terasawa H, Kawai M, Ina S, Hirono S, Uchiyama K, Yamaue H. Improvement of delayed gastric emptying in pylorus-preserving pancreaticoduodenectomy: results of a prospective, randomized, controlled trial. Ann Surg. 2006 Mar;243(3):316-20. doi: 10.1097/01.sla.0000201479.84934.ca. PMID 16495694
- [Background] Tani M, Onishi H, Kinoshita H, Kawai M, Ueno M, Hama T, Uchiyama K, Yamaue H. The evaluation of duct-to-mucosal pancreaticojejunostomy in pancreaticoduodenectomy. World J Surg. 2005 Jan;29(1):76-9. doi: 10.1007/s00268-004-7507-0. PMID 15592915
- [Background] Tani M, Kawai M, Terasawa H, Ueno M, Hama T, Hirono S, Ina S, Uchiyama K, Yamaue H. Complications with reconstruction procedures in pylorus-preserving pancreaticoduodenectomy. World J Surg. 2005 Jul;29(7):881-4. doi: 10.1007/s00268-005-7697-0. PMID 15951940
- [Derived] Busquets J, Martin S, Fabregat J, Secanella L, Pelaez N, Ramos E. Randomized trial of two types of gastrojejunostomy after pancreatoduodenectomy and risk of delayed gastric emptying (PAUDA trial). Br J Surg. 2019 Jan;106(1):46-54. doi: 10.1002/bjs.11023. Epub 2018 Dec 3. PMID 30507039
- [Derived] Tani M, Kawai M, Hirono S, Okada KI, Miyazawa M, Shimizu A, Kitahata Y, Yamaue H. Randomized clinical trial of isolated Roux-en-Y versus conventional reconstruction after pancreaticoduodenectomy. Br J Surg. 2014 Aug;101(9):1084-91. doi: 10.1002/bjs.9544. Epub 2014 Jun 26. PMID 24975853